CLINICAL TRIAL: NCT06715176
Title: Prognostic Utility of TREM-1 Pathway in Predicting Treatment Outcomes in Patients With Grades B and C Periodontitis
Brief Title: TREM-1 Pathway in Predicting Treatment Outcomes in Periodontitis
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Beral Afacan, Assoc. Prof., Aydin Adnan Menderes University
Other Study IDs: TREM-1 pathway
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing; Triiodothyronine

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Unstimulated whole saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Periodontal Health: This group showed PD ≤ 3 mm with BOP < 10 % in the entire mouth as well as no interproximal CAL or radiographic bone loss.
  Interventions: Other: Clinical periodontal measurements at baseline (T0); Other: Saliva collection at baseline (T0)
- Gingivitis: This group exhibited PD ≤ 3 mm with BOP ≥ 30 % in the entire mouth as well as no interproximal CAL or radiographic bone loss.
  Interventions: Other: Clinical periodontal measurements at baseline (T0); Other: Saliva collection at baseline (T0)
- Stage III, Grade B Periodontitis: This group had interproximal CAL ≥ 5 mm along with PD ≥ 6 mm and radiographic bone loss extending to the middle or apical third of the root radiographically at 30 % of the teeth or more. CAL was not caused by trauma-related gingival recession, dental caries extending into the cervical areas of the teeth, endodontic lesions draining through the marginal periodontium, and the distal bone loss in adjacent second molars due to extractions of third molars. They had ≤ 4 teeth lost owing to periodontitis. % of radiographic bone loss/age value was between 0.25 and 1.0.
  Interventions: Other: Clinical periodontal measurements at baseline (T0); Other: Saliva collection at baseline (T0); Other: Scaling and root planing; Other: Clinical periodontal measurements at T1, T3, and T6.; Other: Saliva collection at T1, T3, and T6.
- Stage III, Grade C Periodontitis: This group had interproximal CAL ≥ 5 mm along with PD ≥ 6 mm and radiographic bone loss extending to the middle or apical third of the root radiographically at 30 % of the teeth or more. CAL was not caused by trauma-related gingival recession, dental caries extending into the cervical areas of the teeth, endodontic lesions draining through the marginal periodontium, and the distal bone loss in adjacent second molars due to extractions of third molars. They had ≤ 4 teeth lost owing to periodontitis. % of radiographic bone loss/age were value was higher than 1.0.
  Interventions: Other: Clinical periodontal measurements at baseline (T0); Other: Saliva collection at baseline (T0); Other: Scaling and root planing; Other: Clinical periodontal measurements at T1, T3, and T6.; Other: Saliva collection at T1, T3, and T6.

INTERVENTIONS:
Other: Clinical periodontal measurements at baseline (T0) — Full-mouth clinical periodontal measurements, including PD, CAL, GI, and PI were recorded at 6 sites per tooth, except the third molars, at baseline (T0). A manual periodontal probe was used for PD (millimeters) and CAL (millimeters) measurements; the cemento-enamel junction was used as a reference point for the measurement of CAL.
Other: Saliva collection at baseline (T0) — Unstimulated whole saliva was collected from all participants at baseline (T0). The participants were instructed to refrain from mechanical or chemical oral hygiene practices, eating, drinking, and chewing gum for 2 hours prior to sample collection. Every participant rinsed the mouth with tap water for 2 minutes. Ten minutes after rinsing, they were told to allow the accumulation of the saliva in their mouths and then to drain passively the saliva pool from the lower lip into a steril container for 5 minutes.
Other: Scaling and root planing — Periodontitis patients (grade B and C) underwent a program of non-surgical periodontal therapy consisting of conventional quadrant-based scaling and root planing using ultrasonic instruments and manual periodontal curette over four visits at 1-week intervals. All present teeth were instrumented until the root surface was visually and tactilely clean and smooth. Patients who did not respond to treatment at baseline (T0) received a further round of scaling and root planing at three (T3) months post-therapy in order to eliminate residual pockets.
  Groups: Stage III, Grade B Periodontitis; Stage III, Grade C Periodontitis
Other: Clinical periodontal measurements at T1, T3, and T6. — Full-mouth clinical periodontal measurements were performed for all periodontitis patients (grade B and C) at one (T1), three (T3) and six (T6) months after scaling and root planing.
  Groups: Stage III, Grade B Periodontitis; Stage III, Grade C Periodontitis
Other: Saliva collection at T1, T3, and T6. — Unstimulated whole saliva were collected from all periodontitis patients (grade B and C) at one (T1), three (T3) and six (T6) months after scaling and root planing.
  Groups: Stage III, Grade B Periodontitis; Stage III, Grade C Periodontitis

SUMMARY:
This study investigated modulations in salivary triggering receptor expressed on myeloid cells (TREM)-1, peptidoglycan recognition protein 1 (PGLYRP1) and interleukin (IL)-1β levels between healthy, gingivitis and periodontitis patients, and in response to non-surgical periodontal treatment. Systemically healthy, non-smokers with gingivitis (n=31), stage III periodontitis (grade B: n=34, grade C: n=24) and periodontally-healthy controls (n=34) were recruited. Periodontitis patients (n=45) underwent non-surgical periodontal treatment. Saliva was collected at baseline (T0, all groups), and three times (T1, T3 and T6) post-treatment (periodontitis groups only). Salivary biomarkers and total protein were measured using commercial assays.

DETAILED DESCRIPTION:
Study population and design: For this study, systemically healthy, non-smokers with gingivitis (n = 31), stage III, grade B periodontitis (n = 34), stage III, grade C periodontitis (n = 24), and periodontally healthy controls (n = 34) were recruited at the Department of Periodontology, School of Dentistry, Aydın Adnan Menderes University, Aydın, Turkey.

Clinical examination and saliva collection: All participants were clinically examined at baseline (T0) and whole mouth plaque (PI) and gingival index (GI), probing depth (PD), bleeding on probing (BOP) and clinical attachment loss (CAL) were measured. Prior to clinical examinations, unstimulated whole saliva was collected from all participants at baseline (T0). Additionally, saliva sampling and clinical examinations were performed for all periodontitis patients (grade B and C) one (T1), three (T3) and six (T6) months after non-surgical periodontal treatment.

Non-surgical periodontal treatment protocol: The patients underwent non-surgical periodontal therapy including quadrant-based scaling and root planning (SRP) using ultrasonic instruments and periodontal curettes until the root surfaces were visibly and tactically clean and smooth. All participants were given routine oral hygiene instructions and asked to abstain from any anti-inflammatory drugs, antibiotics, or mouthwashes containing chlorhexidine throughout the study period. At every visit, oral hygiene instructions were reinforced, and the sites that did not respond to treatment at T1 underwent additional re-instrumentation at T3 and T6. While non-surgical treatment efficacy is often reported in terms of mean values of PD reduction and CAL gain, these metrics may not fully capture treatment success or periodontal stability.

Triggering receptor expressed on myeloid cells (TREM)-1, peptidoglycan recognition protein 1 (PGLYRP1) and interleukin (IL)-1β immunoassays and total protein determination: 249 saliva samples were included for the analysis of TREM-1, PGLYRP1 and IL-1β. Levels of those cytokines in saliva were measured by commercial enzyme-linked immunosorbent assays according to manufacturer's instructions. Total protein levels in saliva were measured by the BCA Protein Assay according to the manufacturer's guidelines.

Statistical analysis: Group comparisons were performed with Mann-Whitney, Kruskal-Wallis with Dunn-Bonferroni post-hoc, or Chi-square tests, whenever appropriate. Group comparisons before and after treatment were performed with Friedman with Dunn-Bonferroni post-hoc test. Differences were deemed statistically significant at p ≤0.05.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy
* non-smoker individuals

Exclusion Criteria:

* pregnancies or lactation
* to exposure to antibiotics or any other drugs that were known to affect periodontal conditions over the past 6 months prior to recruitment.
* to receive previous surgical/nonsurgical periodontal treatment during the previous 12-months.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: For this observational study, systemically healthy, non-smokers with gingivitis (n = 31), stage III, grade B periodontitis (n = 34), stage III, grade C periodontitis (n = 24), and periodontally healthy controls (n = 34) were consecutively recruited at the Department of Periodontology, School of Dentistry, Aydın Adnan Menderes University, Aydın, Turkey.
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2016-12-19 (Actual); Primary Completion 2018-01-03 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Salivary TREM-1 level | Change from baseline to one, three and six months after scaling and root planing
  Salivary TREM-1 concentration (pg/ml)
Salivary PGLYRP1 level | Change from baseline to one, three and six months after scaling and root planing
  Salivary PGLYRP1 concentration (ng/ml)
Salivary IL-1β level | Change from baseline to one, three and six months after scaling and root planing
  Salivary IL-1β concentration (pg/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Nagihan Bostanci, Principal Investigator — Karolinska Institutet
Locations (1):
- Aydın Adnan Menderes University, Faculty of Dentistry, Department of Periodontology, Aydin, Turkey (Türkiye)

REFERENCES:
- [Derived] Silbereisen A, Lira-Junior R, Afacan B, Ozturk OV, Emingil G, Bostanci N. TREM-1 Pathway Biomarkers for Classification of Periodontal Diseases and Monitoring of Treatment Response in Grade B and C Periodontitis. J Clin Periodontol. 2025 Sep;52(9):1288-1297. doi: 10.1111/jcpe.14195. Epub 2025 Jun 17. PMID 40528650